CLINICAL TRIAL: NCT04328649
Title: Clinical, Structural and Mechanical Features in Patients With Left Bundle Branch Block: an Observational and Prospective Study.
Brief Title: Clinical, Structural and Mechanical Features in Patients With Left Bundle Branch Block.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Policlinico Casilino ASL RMB (Other)
Responsible Party: Principal Investigator, Leonardo Calò, MD, Professor, FESC, Policlinico Casilino ASL RMB
Other Study IDs: PoliclinicoCasilino
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Left Bundle-Branch Block; Electrocardiographic Pattens; Clinical Features
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical, structural and mechanical features in patients with left bundle branch block.

DETAILED DESCRIPTION:
Left bundle-branch block (LBBB) is an electrocardiographic marker often associated with underlying cardiac disease (such as coronary artery disease, dilated cardiomyopathy, etc) but in some cases it is also found in patients with isolated LBBB defined as "none apparent structural heart disease".

Several investigations in animal and human study have showed a different electroanatomical activation in isolated LBBB when compared to LBBB in heart failure patients mostly due to coronary artery disease. The sequence of endocardial activation through the left ventricle has also proven to be heterogeneous in heart failure occuring at different septal regions. This electrical and mechanical variability seems to be related to location of LBBB block or lesion that could be proximal, distal or diffuse, consequently influencing also electrocardiographic aspects.

These considerations explain and justify the great variability in the proposed "true or typical LBBB" definitions (derived from from Strauss, Perrin and Marican definitions and from Heart Association/American College Cardiology Foundation/ European Society of Cardiology guidelines) but also shift attention to relatively new concept of atypical LBBB definitions with extreme left or right axis deviation and of non specific intraventricular conduction delay defined as a wide QRS (≥110 ms) without the appearance of left and right bundle-branch block. In fact, several investigations have shown that QRS axis deviation is a predictor of unfavorable outcome after cardiac resynchronization therapy and LBBB. The less favorable outcome of cardiac resynchronization therapy candidates with LBBB and left axis deviation seems to be associated to the presence of a shorter activation delay, scar tissue and left ventricular hypertrophy. Moreover, actual LBBB definitions recommended by guidelines in cardiac resynchronization therapy patients differ significantly and only individual ECG criteria (such as electrocardiographic intervals QS or RS in lead V1, notch and no q wave in lead V5, V6, I and avL) seems to be associated to clinical outcome when compared with combining criteria.

Finally, a frequent dyssynchrony of ventricular activation due to LBBB may be responsible for a dyssynchrony-related cardiomyopathy that needs to be identified early and differentiated from other forms of dilated cardiomyopathy through a multiparametric approach such as genetic, clinical data, electrocardiography and cardiac magnetic resonance. In fact, in isolated LBBB undergone cardiac magnetic resonance it was observed a greater left ventricular volumes and lower global left ventricular Ejection Fraction despite the absence of cardiovascular disease as compared with control subject. Despite this, comparison between isolated LBBB and structural heart disease shows a different myocardial mechanism all the more unfavourable the more significant is the presence of underlying myocardial scarring. In the other hand, isolated LBBB, dyssynchrony-related cardiomyopathy and myocardial scarring could present different temporal phase in the clinical history of the same patient and that must be early identified.

The aim of this present large-scale prospective observational study is to evaluate 1) clinical, electrocardiographic and imaging features in a population of patients with typical and atypical LBBB and " non specific intraventricular conduction delay" pattern during a long-term follow up and 2) association among eventual different LBBB patterns (typical, atypical (LBBB and extreme left and/or right axis deviation, fragmentation) and " non specific intraventricular conduction delay " pattern and tissue characterization, mechanical myocardial activation and perfusion. 3) a possible time-related evolution from "non specific intraventricular conduction delay" patterns to typical or atypical LBBB.

ELIGIBILITY:
Inclusion Criteria:

* Every patient with electrocardiographic diagnosis of LBBB admitted to our Cardiology Department and Ambulatory Care Unit
* ECG standard criteria from typical, atypical and NIVCD
* Patients who have given their informed consent in writing.
* Age ≥ 18 years

Exclusion Criteria:

* Age <18 years
* Patients who have not given their informed consent in writing.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In this prospective observational study we consider to enroll patients with LBBB admitted to our Cardiology Department and Ambulatory Care Unit recording different ECG patterns, risk factors, genetic, underlying heart disease, imaging parameters (Echocardiographic and Cardiac Magnetic Resonance) and treatment (either pharmacological or interventional).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Rate of ECG pattern distribution in LBBB patients | 5 years
Rate of underlying structural heart diseases in different LBBB pattern | 5 years
Number of participants with stress induced myocardial ischemia during Stress Magnetic resonance | 5 years
number or participants with late gadolinium enhancement during cardiac magnetic resonance | 5 years
number and of participants with isolated LBBB evolving to dyssynchrony-related cardiomyopathy | 5 years
Number of participants with mechanical dyssynchrony evaluated with Echocardiography | 5 years
  Strain, Strain Rate, intraventricular timing Delay between left ventricular lateral and Septal wall

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akhtari S, Chuang ML, Salton CJ, Berg S, Kissinger KV, Goddu B, O'Donnell CJ, Manning WJ. Effect of isolated left bundle-branch block on biventricular volumes and ejection fraction: a cardiovascular magnetic resonance assessment. J Cardiovasc Magn Reson. 2018 Sep 20;20(1):66. doi: 10.1186/s12968-018-0457-8. PMID 30231875
- [Background] Strik M, Regoli F, Auricchio A, Prinzen F. Electrical and mechanical ventricular activation during left bundle branch block and resynchronization. J Cardiovasc Transl Res. 2012 Apr;5(2):117-26. doi: 10.1007/s12265-012-9351-1. Epub 2012 Feb 7. PMID 22311563
- [Background] Surawicz B, Childers R, Deal BJ, Gettes LS, Bailey JJ, Gorgels A, Hancock EW, Josephson M, Kligfield P, Kors JA, Macfarlane P, Mason JW, Mirvis DM, Okin P, Pahlm O, Rautaharju PM, van Herpen G, Wagner GS, Wellens H; American Heart Association Electrocardiography and Arrhythmias Committee, Council on Clinical Cardiology; American College of Cardiology Foundation; Heart Rhythm Society. AHA/ACCF/HRS recommendations for the standardization and interpretation of the electrocardiogram: part III: intraventricular conduction disturbances: a scientific statement from the American Heart Association Electrocardiography and Arrhythmias Committee, Council on Clinical Cardiology; the American College of Cardiology Foundation; and the Heart Rhythm Society. Endorsed by the International Society for Computerized Electrocardiology. J Am Coll Cardiol. 2009 Mar 17;53(11):976-81. doi: 10.1016/j.jacc.2008.12.013. No abstract available. PMID 19281930
- [Background] European Society of Cardiology (ESC); European Heart Rhythm Association (EHRA); Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE. 2013 ESC guidelines on cardiac pacing and cardiac resynchronization therapy: the task force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Europace. 2013 Aug;15(8):1070-118. doi: 10.1093/europace/eut206. Epub 2013 Jun 24. No abstract available. PMID 23801827
- [Background] Strauss DG, Selvester RH, Wagner GS. Defining left bundle branch block in the era of cardiac resynchronization therapy. Am J Cardiol. 2011 Mar 15;107(6):927-34. doi: 10.1016/j.amjcard.2010.11.010. PMID 21376930
- [Background] Padanilam BJ, Morris KE, Olson JA, Rippy JS, Walsh MN, Subramanian N, Vidal A, Prystowsky EN, Steinberg LA. The surface electrocardiogram predicts risk of heart block during right heart catheterization in patients with preexisting left bundle branch block: implications for the definition of complete left bundle branch block. J Cardiovasc Electrophysiol. 2010 Jul;21(7):781-5. doi: 10.1111/j.1540-8167.2009.01714.x. Epub 2010 Feb 1. PMID 20132380
- [Background] Kisiel R, Fijorek K, Moskal P, Kukla P, Pavlinec C, Stec J, Czarnecka D, Jastrzebski M. True left bundle branch block and long-term mortality in cardiac resynchronisation therapy patients. Kardiol Pol. 2019;77(3):371-379. doi: 10.5603/KP.a2019.0032. Epub 2019 Feb 25. PMID 30799545
- [Background] Eschalier R, Ploux S, Ritter P, Haissaguerre M, Ellenbogen KA, Bordachar P. Nonspecific intraventricular conduction delay: Definitions, prognosis, and implications for cardiac resynchronization therapy. Heart Rhythm. 2015 May;12(5):1071-9. doi: 10.1016/j.hrthm.2015.01.023. Epub 2015 Jan 19. PMID 25614250
- [Background] Storkas HS, Hansen TF, Tahri JB, Lauridsen TK, Olsen FJ, Borgquist R, Vinther M, Lindhardt TB, Bruun NE, Sogaard P, Risum N. Left axis deviation in patients with left bundle branch block is a marker of myocardial disease associated with poor response to cardiac resynchronization therapy. J Electrocardiol. 2020 Nov-Dec;63:147-152. doi: 10.1016/j.jelectrocard.2019.04.007. Epub 2019 Apr 5. PMID 31003852
- [Background] van Stipdonk AMW, Hoogland R, Ter Horst I, Kloosterman M, Vanbelle S, Crijns HJGM, Prinzen FW, Meine M, Maass AH, Vernooy K. Evaluating Electrocardiography-Based Identification of Cardiac Resynchronization Therapy Responders Beyond Current Left Bundle Branch Block Definitions. JACC Clin Electrophysiol. 2020 Feb;6(2):193-203. doi: 10.1016/j.jacep.2019.10.009. Epub 2019 Nov 27. PMID 32081223
- [Background] Sanna GD, Merlo M, Moccia E, Fabris E, Masia SL, Finocchiaro G, Parodi G, Sinagra G. Left bundle branch block-induced cardiomyopathy: a diagnostic proposal for a poorly explored pathological entity. Int J Cardiol. 2020 Jan 15;299:199-205. doi: 10.1016/j.ijcard.2019.06.008. Epub 2019 Jun 4. PMID 31186131
- [Background] Strauss DG, Selvester RH. The QRS complex--a biomarker that "images" the heart: QRS scores to quantify myocardial scar in the presence of normal and abnormal ventricular conduction. J Electrocardiol. 2009 Jan-Feb;42(1):85-96. doi: 10.1016/j.jelectrocard.2008.07.011. Epub 2008 Sep 13. No abstract available. PMID 18790501